CLINICAL TRIAL: NCT00957814
Title: Impact of Nutritional Orientations on Adherence to Diet and Relation to Nutritional, Clinical and Life Quality Parameters of Heart Failure Outpatients
Brief Title: Nutritional Orientations and Adherence, Nutritional Status, Clinical and Life Quality Parameters of Heart Failure (HF) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ingrid Dalira Schweigert, Dr., Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UFRGS and HCPA 14741
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Nutrition; Heart Failure
Keywords: nutritional education; diet adherence; nutritional knowledge; life quality; nutritional status; impact of nutritional orientations by a systematic education program applied to outpatients with HF, in comparison to patients in a conventional treatment.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): Usual care with medical and nursing staff
  Interventions: Behavioral: Nutritional education
- Intervention (Experimental): Usual care with medical and nursing staff and additional nutritional guidance about diet and its relationship with disease, sources of nutrients, and reduction of dietary sodium and fats. Enforcement of the nutritional guidance was performed after 4 weeks.
  Interventions: Behavioral: Nutritional education

INTERVENTIONS:
Behavioral: Nutritional education — Systematic nutritional orientation program

SUMMARY:
The nutritional systematic orientations in outpatients with heart failure throughout 1 year in comparison to conventional treatment is estimated to lead to higher nutritional treatment adherence and improved nutritional status, clinical and life quality parameters.

DETAILED DESCRIPTION:
To evaluate the impact of systematic nutritional orientation on adherence to diet and relation to clinical, life quality and nutritional knowledge parameters in heart failure outpatients.

* To evaluate the impact of systematic nutritional orientation on nutritional status;
* To evaluate the impact of nutritional systematic orientation on dietary patterns
* To evaluate the impact of systematic nutritional orientation on clinical and biochemical parameters
* To evaluate the impact of nutritional systematic orientation on life quality
* To evaluate the impact of nutritional systematic orientation on nutritional knowledge

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Outpatients from the HF Ambulatory (HCPA)
* Functional class I and II (NYHA)

Exclusion Criteria:

* Outpatient who had received any orientation from a nutritionist in the last 6 months
* Outpatients which has not received nursing orientation in the ambulatory,
* Patients from other NYHA class
* Non alphabetized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Diet adherence | 1 year

SECONDARY OUTCOMES:
Knowledge about nutrition, nutritional status, biochemical parameters and life quality | 1 year